CLINICAL TRIAL: NCT02209467
Title: Balance and Falls in Multiple Sclerosis: Intervention and Perceptions From Patients and Next of Kins
Brief Title: Balance and Falls in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro County Council (Other Government)
Responsible Party: Principal Investigator, Anette Forsberg, PhD, PhD, lecturer, Örebro County Council
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Researchweb 153691
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Multiple Sclerosis
Keywords: walking; postural balance; falls
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group balance training late start (No Intervention): Participants randomized to late start act as No intervention group during the study period.
- Group balance training early start (Experimental): Group balance training focusing on core stability exercises 2 times per week for 7 weeks and 2 home training sessions per weeks.
  Interventions: Other: Group balance training

INTERVENTIONS:
Other: Group balance training — Group balance training 60 minutes 2 times per week plus 3-5 home exercises 2 times/week. Exercises focus om core stability in sitting, standing and lying.
  Arms: Group balance training early start

SUMMARY:
The study hypothesis is that for people with moderate to severe multiple sclerosis postural balance and walking improve and the risk of accidental falls are reduced after participating in a specific training intervention of 7 weeks. The hypothesis is also the the effect remain a further 7 weeks post training.

Multiple Sclerosis (MS) is disease affecting the central nervous system. Walking and postural balance are often affected early in the course of the disease. The risk of falls is large. Many persons with MS have decreased trunk stability compared to healthy persons . In an earlier study including people with mild to moderate MS we found that a period of core stability exercises reduced the risk of falls. In this study the training concept will be applied for persons with more severe walking limitations.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed multiple sclerosis
* Expanded Disability Scale Score of 5-6.5
* walking speed of less than 0.8 m/s as tested on a 10 meter walking test

Exclusion Criteria:

* Ongoing relapse
* Cognitive or language difficulties that prohibit participating in the intervention or performing the outcome measures
* Change in specific MS medication during the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Berg Balance Scale at 8 weeks | baseline, 8 weeks

SECONDARY OUTCOMES:
Change from baseline in 10 repetitions Sit to stand test at 15 weeks | baseline, 15 weeks
Change from baseline in Trunk Impairment scale at 8 weeks | baseline, 8 weeks
Change from baseline in the Trunk Impairment Scale at 15 weeks | baseline, 15 weeks
Change from baseline in the 10 repetition Si to stand test at 8 weeks | baseline, 8 weeks
Change from baseline in the Berg Balance scale at 15 weeks | baseline, 15 weeks
Change from baseline on the Timed Up and Go test at 8 weeks | baseline, 8 weeks
Change from baseline on the Timed Up and Go test at 15 weeks | baseline, 15 weeks
Change from baseline on the10 meter walking test at 8 weeks | baseline, 8 weeks
Change from baseline on the 10 meter walking test at 15 weks | baseline, 15 weeks
Change from baseline on the 2 minutes walking test at 8 weeks | baseline, 8 weeks
Change from baseline on the 2 minutes walking test at 15 weeks | baseline, 15 weeks
Change from baseline in postural sway at 8 weeks | baseline, 8 weeks
Change from baseline in postural sway at 15 weeks | baseline, 15 weeks
  postural sway in standing on the floor is assessed
Change from baseline on the Falls-Efficacy scale at 8 weeks | baseline, 8 weeks
Change from baseline on the Falls Efficacy scale at 15 weeks | baseline, 15 weeks
Change from baseline on the Fatigue Scale for Motor and Cognitive functions at 8 weeks | baseline, 8 weeks
Change from baseline on the Fatigue Scale for Motor and Cognitive functions at 15 weeks | baseline, 15 weeks
Change from baseline on the MS Walking Scale-12 at 8 weeks | baseline, 8 weeks
Change from baseline on the MS Walking scale-12 at 15 weeks | baseline, 15 weeks
The number of falls and accidental falls | from baseline to 15 weeks
  the number of falls and accidental falls are noted by the participant in a study-specific falls diary.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Carling, MSc, Principal Investigator — Centre for Health Care Sciences, Örebro County Council; Anette Forsberg, PhD, Study Chair — Family Medicine Research Centre, Örebro County Council; Ylva Nilsagård, PhD, Study Director — Centre for Health Care Sciences, Örebro County Council
Locations (7):
- Sweden (7):
  - Neurorehab Mälarsjukhuset, Eskilstuna
  - Physiotherapy department Gävle hospital, Gävle
  - Rehab unit Karlskoga hospital, Karlskoga
  - Primary Health Care, Linköping
  - Nyköping hospital, Nyköping
  - Physiotherapy department University hospital, Örebro
  - Rehab unit Västerås hospital, Västerås

REFERENCES:
- [Background] Nilsagard YE, von Koch LK, Nilsson M, Forsberg AS. Balance exercise program reduced falls in people with multiple sclerosis: a single-group, pretest-posttest trial. Arch Phys Med Rehabil. 2014 Dec;95(12):2428-34. doi: 10.1016/j.apmr.2014.06.016. Epub 2014 Jul 6. PMID 25004466